CLINICAL TRIAL: NCT04252144
Title: Study of Dietary Patterns and Food Diversity in Russian GERD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Collaborators: Russian Science Foundation (Other)
Responsible Party: Principal Investigator, Vasily Isakov, MD, PhD, Professor, AGAF, Russian Academy of Medical Sciences
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 19-76-30014 GERD
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Gastroesophageal; Reflux With Esophagitis; Gastroesophageal Reflux; GERD; Heartburn; Non-erosive Reflux Disease; Esophagitis
Keywords: food diversity; dietary pattern; healthy eating pattern; oesophagitis; GERD
MeSH Terms: conditions — Esophagitis, Peptic; Gastroesophageal Reflux; Heartburn; Non-Erosive Reflux Disease; Esophagitis | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Dietary assessment with the use of computer-based food frequency questionnaire will be performed to patients with established diagnosis of gastroesophageal reflux disease in comparison to the representatives of a control group (without the disease).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GERD (Experimental): Patients with verified gastroesophageal reflux disease
  Interventions: Procedure: Dietary assessment
- Contol (Other): Mostly healthy subjects who have no symptoms and other manifestations of gastroesophageal reflux disease by complex examination
  Interventions: Procedure: Dietary assessment

INTERVENTIONS:
Procedure: Dietary assessment — Dietary assessment is not within standards of care for patients with gastroesophageal reflux disease in Russia. Subjects enrolled to the study are to be interviewed on most common foods consumption in terms of frequency of use and sizes of portions.
  Other Names: Food frequency questionnaire

SUMMARY:
The aim of the study is to assess food diversity and dietary patterns in Russian GERD patients

DETAILED DESCRIPTION:
The study of dietary patterns may provide complex vision of an association between consumption of specific foods, or groups of food products and manifestations of gastroesophageal reflux disease (symptoms: heartburn and acid regurgitation; endoscopic findings - oesophagitis). Only limited data on this matter are published to the moment and they predominantly concerns outcomes of gastroesophageal reflux disease (oesophageal adenocarcinoma or Barrett's oesophagus). Taking into the consideration that earlier studies found significant differences in consumption of nutrients in different world regions, new data on food patterns of dietary patterns in Russian GERD patients could partly fill in the gap of knowledge on this particular matter.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate (signed the informed consent form);
* willingness to follow all the required procedures;

Exclusion Criteria:

* Pregnant or breast-feeding females;
* Neoplasms, current or by the medical history (except local skin cancer successfully treated);
* History of chest or abdominal surgery, except appendectomy and cholecistectomy (in case when no consequences of these operations like adhesive disease of the abdominal cavity are present);
* Co-morbid conditions which can influence or mask the symptoms of GERD (including, but not limited to: ischaemic heart disease, severe pulmonary disease, severe depression or anxiety, etc);
* the use of concomitant medications that may influence on the symptoms or other manifestations of gastroesophageal reflux disease: NSAIDs, corticosteroids (except topic ones for no longer than 2 weeks), any medications directly influencing mood and function of central nervous system (antidepressants, anxiolytics, anti-anxiety agents, anticonvulsant etc) at the moment of enrolment and during a 2 half-life period of the certain drug;
* the use of medications that influence gastric secretion at the time of enrolment and during 2 week before it;
* any condition of the patient which makes the participation of the patient in the study unreasonable or put him at risk of the condition's exacerbation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
grains consumption diversity | a month
  Mean number of different types of grains consumed in form of different foods or food products a month during 12-months period
meat consumption diversity | a month
  Mean number of different types of meat consumed in form of different foods or food products a month during 12-months period
poultry consumption diversity | a month
  Mean number of different types of poultry consumed in form of different foods or food products a month during 12-months period
fish consumption diversity | a month
  Mean number of different types of fish consumed in form of different foods or food products a month during 12-months period
flour consumption diversity | a month
  Mean number of different types of flours consumed in form of different foods or food products a month during 12-months period
vegetables consumption diversity | a month
  Mean number of different types of vegetables consumed as is or in the form of different foods or food products
Fruits consumption diversity | a month
  Mean number of different types of fruits consumed as is or in the form of different foods or food products
Fats consumption diversity | a month
  Mean number of different types of fats consumed in the form of different foods or food products a month by 12 month period

SECONDARY OUTCOMES:
GERD-associated dietary pattern | a year
  complex of nutrients and/or foods (food products) which correlates with presence of GERD. The correlation coefficients for each food item is range in the order of significance and direction of the relationship and in accordance to the amount of the product consumed, than is formed to the integral mean.

CONTACTS AND LOCATIONS:
Overall Officials: Vasily Isakov, MD, PhD, Professor, AGAF, Study Chair — FRC nutrition and biotechnology; Sergey Morozov, MD, PhD, Principal Investigator — FRC Nutrition and Biotechnology
Locations (1):
- Gastroenterology and Hepatology, FRC Nutrition and Biotechnology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Study data may be shared by request after study completion, except subjects' personal (identification) information
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the study completion, available for 2 years
Access Criteria: By request
URL: http://ion.ru